CLINICAL TRIAL: NCT04883853
Title: A Newly Modified Technique for Levator Muscle Tucking in Blepharoptosis Surgery: An Egyptian Tertiary Center Study
Acronym: Lidtucking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Mild Ptosis; Moderate Ptosis
Keywords: Ptosis, plication, levator muscle, tucking.
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mild -Moderate Ptosis with good levator function (more than 8 mm) (Experimental): The upper eyelid crease was marked for the incision site, up to 5-7 mm from the lid margin, guided by the fellow eyelid crease position. The skin incision was done and the orbicularis occuli muscle was dissected to the tarsus. The anterior surface of the tarsal plate was then identified with the aponeurosis at its insertion, the orbital septum was then opened with a resultant fat prolapse, and the levator aponeurosis exposed until Whitnall's ligament. Three double-armed 5/0 polyester white braided, non-absorbable sutures, with spatulated needle 1/4 circle (Astralen, Assut Medical Sàrl, Pully-Lausanne, Switzerland) were passed between the levator aponeurosis near Whitnall's ligament and the anterior surface of the tarsus in a mattress form
  Interventions: Procedure: Mild _moderate Ptosis tucking

INTERVENTIONS:
Procedure: Mild _moderate Ptosis tucking — A modified levator muscle tucking procedure.The level of sutures was determined according to the levator muscle function and the desired eyelid height. The middle (main) suture was taken first at the level of the medial part of the pupil and was tightened to keep the lid height at the superior limbus and the other two sutures (medial and lateral) were then adjusted. A spindle-shaped, horizontal part of the levator aponeurosis (2.5-3 mm wide and 0.5 mm deep) was excised at the site of insertion into the tarsus before tightening the central suture to induce strong fibrosis and adhesion between the tucked levator aponeurosis and the tarsus

SUMMARY:
Mild to moderate blepharoptosis with good levator function is usually corrected by levator muscle resection or advancement with their modifications with high success rate. Levator plication technique has been strongly suggested in patients with mild to moderate ptosis, advocated by its simple and rapid recovery. Its drawback is a high recurrence rate.

We suggest a modified tucking technique that improves the force of eyelid elevation with preserved normal anatomy of Muller's muscle and conjunctiva with less disturbance to the Levator muscle aponeurosis. It is a short procedure, less complications with good aesthetic results and high patient's satisfaction.

DETAILED DESCRIPTION:
A prospective single-centre study enrolling 180 patients with blepharoptosis at Ain Shams University Hospitals from March 2017 to February 2019. Patients of unilateral or bilateral mild to moderate ptosis with good levator function (more than 8 mm) were included. Those with severe, traumatic, recurrent, mechanical ptosis, Marcus-Gunn jaw winking syndrome, third nerve palsy, absent Bell's phenomenon, or abnormal ocular motility were excluded. The follow-up was at one week, one month, three months, six months, and one year visits. Functional outcome was assessed by analysis of the upper eyelid margin position in relation to the superior limbus and classified as very good (2 mm), good (2-4 mm), poor (5 mm) and preoperative to postoperative difference in marginal reflex distance (MRD). The aesthetic outcome was assessed in the form of symmetry of eyelid height, lid contour, lid crease presence, and degree of patient's postoperative satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Mild _moderate blepharoptosis

Exclusion Criteria:

* severe, traumatic, recurrent, or mechanical ptosis, third nerve palsy, Marcus-Gunn jaw winking syndrome, abnormal ocular motility, and absent Bell's phenomenon

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
post-operative marginal reflex distance | first day postoperative
  Distance between upper lid margin and pen torch reflex

SECONDARY OUTCOMES:
upper eyelid margin position | first day postoperative
  margin position in relation to the superior limbus in the digital photos

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Ahmed, M.D,FRCS, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of medicine Ain Shams University, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04883853/Prot_SAP_000.pdf